CLINICAL TRIAL: NCT04265209
Title: Non-inferiority Study of the Molecular Imaging of Dopamine Transporters Using [123I]-FP/CIT-SPECT and [18F] LBT-999-PET to Distinguish Between Parkinson's Disease and Essential Tremor.
Brief Title: [18F] LBT-999 PET Compared to [123I]-FP/CIT SPECT to Distinguish Between Parkinson's Diseases and Essential Tremor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZX-2018-LBT999-DATTEP-3
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPECT and PET (Other): [123I]-FP-CIT SPECT imaging procedure first, then [18F] LBT-999 PET Imaging procedure
  Interventions: Drug: SPECT; Drug: PET
- PET and SPECT (Other): [18F] LBT-999 PET imaging procedure first, then [123I]-FP-CIT SPECT imaging procedure
  Interventions: Drug: SPECT; Drug: PET

INTERVENTIONS:
Drug: SPECT — [123I]-FP-CIT SPECT imaging procedure
Drug: PET — [18F] LBT-999 PET imaging procedure

SUMMARY:
Clinical study to demonstrate an at least equivalent performance of a new PET molecular Imaging radiopharmaceutical named [18F] LBT-999 in brain imaging compared to the SPECT reference method named [123I]-FP-CIT to establish the differential diagnosis between Parkinson's Disease and Essential Tremor.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 to 80 (male or female)
* Patients:

  * suffering from an essential tremor as defined by Elble's criteria from 2000 (excluding head tremor in decubitus and compatible with the study by the investigator)
  * or with Parkinson's disease as defined by the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB)
* Patients with clinical symptoms dated more than 18 months ago
* Women of childbearing potential who must have effective contraception at baseline and up to 30 days after the last administration of the radiopharmaceutical (investigational medicinal product or comparator)
* Patients affiliated with or receiving a social security scheme
* Patients who have been fully informed about the organization of the research and who have signed their informed consent

Exclusion Criteria:

* Patients with atypical non-idiopathic Parkinson's syndrome (multi system atrophy, progressive supranuclear palsy, etc.)
* Patients treated with deep brain stimulation
* Patients with functional psychogenic movements
* Patients with severe and progressive psychiatric disorders
* Patients with disabling dyskinesia or essential tremor that are incompatible with imaging studies
* Patients who have had an ionizing radiation examination on the brain within the last 3 months
* Individuals with a contraindication to PET or SPECT imaging:

  * Patients with claustrophobia
  * Patients refusing to be informed in case of abnormalities detected during imaging tests
  * Patients treated with amphetamines, benzatropine, amfebutamone, cocaine, mazindol, methylphenidate, phentermine or sertraline
  * Individuals with a known allergy to the active substance or one of the excipients of the product under investigation or to the reference product or to or to thyroid treatment
* Woman of childbearing age without effective contraception in the opinion of the investigator
* Any other serious unstabilized chronic condition deemed incompatible with the study by the investigator
* Patients unable to sign the informed consent
* Patients participating in a protocol or in a period of exclusion from a protocol
* Patients who received compensation of more than 6000 € in the last 12 months prior to enrollment in clinical studies
* Patients in a period of exclusion from the national volunteer database during which they cannot participate in another clinical study
* Patients not affiliated with a social security scheme
* Patients refusing to participate
* Individuals referred to in articles L. 1121-5 to L. 1121-8 and L1122-2 of the French Public Health Code

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity by visual analysis | The independent review committee will analyse the PET and SPECT images blindly. These analyses will be done by batch of 25 patients. Outcome will be assessed at the end of the study, an average of 2 years after first patient in.
  Sensitivity and specificity of each imaging method on the diagnosis of normal or pathological examination on the visual analysis by 5 independent readers interpreting a minimum of 200 [123I]-FP/CIT SPECT per year, without knowing the clinical diagnosis.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Hôpital Avicenne, Bobigny
  - CHU Bordeaux, Bordeaux
  - Centre Jean PERRIN / Hôpital Gabriel Montpied (CHU), Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CLCC Georges-François Leclerc C.G.F.L, Dijon
  - Hôpital Roger Salengro (CHRU de Lille), Lille
  - Hospices Civils de Lyon, Lyon
  - CHU La Timone, Marseille
  - Hôpital Brabois / Hôpital Central (CHRU Nancy), Nancy
  - Hôpital Laennec (CHU Nantes), Nantes
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - CHU La Pitié Salpêtrière, Paris
  - Centre Eugène Marquis / CHU Pontchaillou, Rennes
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital Pierre Paul Riquet - Purpan (CHU), Toulouse
  - CHRU Hôpital Bretonneau, Tours